CLINICAL TRIAL: NCT03762213
Title: Audio-Visual Relaxation Technology for Pediatric Amplified Musculoskeletal Pain Syndrome: A Pilot Randomized Controlled Trial
Brief Title: Audio-Visual Relaxation Technology for Pediatric Amplified Musculoskeletal Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13135
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Amplified Musculoskeletal Pain Syndrome; Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes
MeSH Terms: conditions — Chronic Pain; Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: The investigators propose a parallel-group pilot randomized controlled trial with a stratified block randomization and an equal allocation ratio of 1:1. The participants will be randomly allocated to Group A (VR/intervention group) or Group B (iPad/control group). The relaxation session will last for 10 minutes in each group using the same application Happy Place (© Mimerse) played on VR headsets (Oculus GO) versus iPad (Apple Inc. Cupertino CA). The randomization will be stratified on the basis of pain score on the day of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Oculus GO VR HMD, application Happy Place (© Mimerse) (Experimental): Oculus GO is a stand-alone, consumer-grade, virtual reality head-mounted display (HMD). The HMD is placed on the head of the user blocking off the surrounding environment. The visuals and audio are relayed through the HMD in a virtual space.Happy Place (© Mimerse) is a publicly available application with an explicit intent to be used for chronic pain patients. It has the critical elements of VR, namely immersion and interactivity.
  Immersion: The scene is a serene lakeside campground with guided relaxation and soothing music. The application intends to promote positive effects such as calmness and feeling of wonder.
  Interactivity: Happy Place uses an innovative 'gaze-based interaction' with the virtual world. Around 50 'gaze objects' are placed around the scene and gazing at them would trigger an event.
  The entire duration of the experience will be kept at 10 minutes.
  Interventions: Device: Oculus GO VR HMD, application Happy Place (© Mimerse)
- iPad, application Happy Place (© Mimerse) (Placebo Comparator): An iPad with earphones (Apple Inc. Cupertino CA) will be used for controls. The participants in control group will watch the same content for the same duration on an iPad screen (flat version of Happy Place). This experience will be different from the intervention group in two ways: first, lack of an immersive environment, and second, lack of interactivity with the environment.
  Interventions: Device: iPad, application Happy Place (© Mimerse)

INTERVENTIONS:
Device: Oculus GO VR HMD, application Happy Place (© Mimerse) — The Entertainment Software Rating Board (ESRB) has rated Happy Place as 'E' ('Everyone' or content suitable for all ages).
  Arms: Oculus GO VR HMD, application Happy Place (© Mimerse)
Device: iPad, application Happy Place (© Mimerse) — The Entertainment Software Rating Board (ESRB) has rated Happy Place as 'E' ('Everyone' or content suitable for all ages).
  Arms: iPad, application Happy Place (© Mimerse)

SUMMARY:
A pilot randomized controlled trial to assess feasibility, acceptability and generate outcome domains for a future RCT testing the efficacy of immersive virtual reality on pain intensity in pediatric amplified musculoskeletal pain syndrome.

DETAILED DESCRIPTION:
Adolescents with amplified musculoskeletal pain syndrome (AMPS) are invited to take part in this research project that studies two different audio-visual relaxation technologies in reducing amplified musculoskeletal pain. In addition, the investigators are interested in studying if they have an effect on some of the ways adolescents think about their pain and cope with it. Both of these technologies provide the user with a similar natural environment designed to have a calming effect, along with guided relaxation and soothing music. The adolescents will be assigned to use one of these for a total duration of about 10 minutes. Pain related outcomes including pain intensity, pain catastrophizing and self-efficacy to manage pain will be collected before and after the relaxation session.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of AMPS, including CRPS, or localized or diffuse amplified pain syndrome as determined by the primary pediatric rheumatologist and coded in EMR.
2. Informed consent for caregivers and child assent for participants.

Exclusion Criteria:

1. An underlying organic cause can explain the pain including inflammatory, infectious, traumatic or malignant etiologies as determined by the primary pediatric rheumatologist.
2. Participant or caregiver report of any history of motion sickness, underlying epilepsy, severe headaches in the participant or other conditions where the use of visual exposures to stimuli is contraindicated.
3. Inability to report a pain score and/or incapacity to give assent due to intellectual deficit.
4. Blindness.
5. Non-English-speaking subjects will be excluded due to the unavailability of the content of the VR application used in this study in languages other than English.
6. Any other condition that the investigators think can compromise the integrity of the study or subject safety.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor E Davis, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oculus GO VR HMD, Application Happy Place (© Mimerse): Oculus GO is a stand-alone, consumer-grade, virtual reality head-mounted display (HMD). The HMD is placed on the head of the user blocking off the surrounding environment. The visuals and audio are relayed through the HMD in a virtual space.Happy Place (© Mimerse) is a publicly available application with an explicit intent to be used for chronic pain patients. It has the critical elements of VR, namely immersion and interactivity.
  Immersion: The scene is a serene lakeside campground with guided relaxation and soothing music. The application intends to promote positive effects such as calmness and feeling of wonder.
  Interactivity: Happy Place uses an innovative 'gaze-based interaction' with the virtual world. Around 50 'gaze objects' are placed around the scene and gazing at them would trigger an event.
  The entire duration of the experience will be kept at 10 minutes.
  Oculus GO VR HMD, application Happy Place (© Mimerse): The Entertainment Software Rating Board (ESRB) has rated Happy Place as 'E' ('Everyone' or content suitable for all ages).
Period: Overall Study
Arm/Group | Oculus GO VR HMD, Application Happy Place (© Mimerse) | iPad, Application Happy Place (© Mimerse)
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oculus GO VR HMD, Application Happy Place (© Mimerse) | iPad, Application Happy Place (© Mimerse) | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.1) | 15.4 (1.5) | 15.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 10 | 22
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change in Pain Intensity Reported on Visual Analog Scale (VAS)
Description: The VAS is a self-reported quantitative measure of pain intensity used commonly in clinical practice as well as in pain research. The VAS is a straight horizontal line of fixed length, usually 0 mm to 100 mm where 0 denotes 'no pain' and 100 denotes 'pain as bad as it could possibly be'. The participant marks a point on the line that they feel represents the perception of their current pain. The VAS score is then determined by measuring in millimeters from the left-hand end of the line to the point that the participant marks. The primary outcome measure is is the mean change in VAS from 5 minutes before the relaxation session to 5 minutes after the session.
Time Frame: VAS will be administered at 5 minutes before the relaxation session, 5 minutes after the session and then at day 2 after the session in both groups.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oculus GO VR HMD, Application Happy Place (© Mimerse) | iPad, Application Happy Place (© Mimerse)
Number analyzed (Participants) | 16 | 14
units on a scale | -14.9 [-22.9 to -6.9] | -9.6 [-14.3 to -4.9]

2. Secondary Outcome: Mean Change in Pain Catastrophizing Reported on Pain Catastrophizing Scale - Child (PCS-C)
Description: The Pain Catastrophizing Scale -Child (PCS-C) is an adaptation of the Pain Catastrophizing Scale with established construct and predictive validity in 8-16 years old subjects. It is a self-report measure which includes 13 items about the thoughts and feelings experienced when a child is in pain. Respondents use a 5-point rating scale (where 0 = never to 4 = always), to indicate how often they experience each thought or feeling. The total score for the PCS equals 52, with a score above 24 indicating a high score. The lowest score can be 0. Higher score represents worse outcome. PCS-C scale has three sub-scales namely, rumination, magnification, and helplessness. The investigators will not assess the sub-scales as a part of this study. The outcome measure will be reported as the mean difference in post-intervention score (assessed 5 minutes after the session) minus pre-intervention score (assessed 5 minuets before the session) for both groups with the 95% confidence interval.
Time Frame: PCS-C will be administered at 5 minutes before the relaxation session, 5 minutes after the session and day 2 after the study.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oculus GO VR HMD, Application Happy Place (© Mimerse) | iPad, Application Happy Place (© Mimerse)
Number analyzed (Participants) | 16 | 14
units on a scale | -2.0 [-4.1 to -0.1] | -2.9 [-5.9 to -0.2]

3. Other Pre Specified Outcome: Mean Change in Self-efficacy to Manage Pain Reported on Self-Efficacy Scale for Child Functioning (SES-C)
Description: The Self-Efficacy Scale for Child Functioning (SES-C) is a reliable and validated self-efficacy measure for children 9-18 years of age with chronic pain. The child version has established psychometric properties, excellent reliability and strong evidence for construct validity. It consists of 7 Likert scale questions with a range from very sure (=1) to very unsure (=5). The lowest score can be 7, which reflects highest self-efficacy to manage pain, and the highest score can be 35, which corresponds to lowest self-efficacy to manage pain. Higher score represents worse outcome. It has no sub-scales. The outcome measure will be reported as the mean difference in post-intervention score (assessed 5 minutes after the session) minus pre-intervention score (assessed 5 minuets before the session) for both groups with the 95% confidence interval.
Time Frame: SES-C will be administered at 5 minutes before the relaxation session, 5 minutes after the session and then at day 2 after the session in both groups.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oculus GO VR HMD, Application Happy Place (© Mimerse) | iPad, Application Happy Place (© Mimerse)
Number analyzed (Participants) | 16 | 14
units on a scale | -0.7 [-1.2 to -0.1] | -2.4 [-4.6 to -0.2]

ADVERSE EVENTS:
Time Frame: 2 days after the session for each participant.
Arm/Group | Oculus GO VR HMD, Application Happy Place (© Mimerse) | iPad, Application Happy Place (© Mimerse)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 9/16 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oculus GO VR HMD, Application Happy Place (© Mimerse) (N=16) | iPad, Application Happy Place (© Mimerse) (N=14)
Dizziness (General disorders) | 3 | 1 — Moderate dizziness >30 on a scale of 0-100
Nausea (General disorders) | 2 | 2 — Moderate nausea >30 on a scale of 0-100
Headache (General disorders) | 4 | 2 — Moderate headache >30 on a scale of 0-100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03762213/Prot_SAP_001.pdf